CLINICAL TRIAL: NCT00003519
Title: Phase III Study of Adriamycin/Taxotere Versus Adriamycin/Cytoxan for the Adjuvant Treatment of Node Positive or High Risk Node Negative Breast Cancer
Brief Title: Combination Chemotherapy in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); North Central Cancer Treatment Group (Network); Cancer and Leukemia Group B (Network)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066563; E2197; CLB-49802; NCCTG-E2197; SWOG-E2197
Record Dates: First submitted 1999-11-01; First posted 2004-08-26 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two combination chemotherapy regimens in treating women with breast cancer who have undergone surgery to remove the tumor.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether doxorubicin/docetaxel (DD) will improve disease-free survival and overall survival when compared to doxorubicin/cyclophosphamide (DC) in women with lymph node positive (1-3 positive nodes) or high risk lymph node negative breast cancer. II. Compare the toxicity of DD to DC in this patient population.

OUTLINE: This is a randomized study. Patients are stratified by node status (positive vs negative), menopause status (pre- vs post), estrogen receptor (ER) status/progesterone receptor (PR) status (ER/PR unknown vs ER+/PR+ vs ER+/PR- vs ER-/PR+ vs ER-/PR-). Patients in arm I receive doxorubicin IV plus docetaxel IV over 1 hour every 3 weeks for 4 treatment courses. Patients in arm II receive doxorubicin IV plus cyclophosphamide IV every 3 weeks for 4 treatment courses. All patients who are estrogen receptor or progesterone receptor positive receive oral tamoxifen daily for 5 years following chemotherapy. Some patients may also receive radiotherapy following chemotherapy. Patients are followed every 3 months if patient is less than 2 years from study entry; every 6 months if patient is 2-5 years from study entry; and every 12 months if patient is greater than 5 years from study entry.

PROJECTED ACCRUAL: Approximately 2778 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed resectable adenocarcinoma of the breast Histologically positive lymph nodes (1 to 3) OR Lymph node negative and high risk disease Tumor greater than 1.0 cm diameter May have undergone an axillary dissection with at least 6 nodes removed and examined or a sentinel node biopsy Patients who are positive by sentinel node biopsy will receive an axillary dissection No locally advanced or inflammatory or metastatic breast cancer Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Adequate hepatic function Bilirubin no greater than upper limit of normal Renal: Adequate renal function Cardiovascular: Adequate cardiac function Normal MUGA or echocardiogram Other: Not pregnant or nursing Fertile patients must use effective barrier method contraception At least 5 years since prior invasive malignancies, except basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for this malignancy Endocrine therapy: No concurrent tamoxifen Up to 4 weeks of tamoxifen treatment for this malignancy allowed Radiotherapy: No prior radiotherapy for this malignancy Prior radiotherapy to the breast for ductal carcinoma in situ allowed Surgery: Tumor should be removed by either a modified radical mastectomy and/or a segmental mastectomy plus axillary lymph node dissection or sentinel node biopsy before beginning treatment on protocol No greater than 84 days since last surgical procedure that constitutes or completes definitive surgical therapy (mastectomy; axillary dissection/sentinel node biopsy; or resection of primary site to obtain a negative margin

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2778 (Estimated)
Dates: Start 1998-08-20 (Actual); Primary Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori J. Goldstein, MD, Study Chair — Fox Chase Cancer Center; Silvana Martino, DO, Study Chair — Van Nuys Breast Center; Edith A. Perez, MD, Study Chair — Mayo Clinic; Larry Norton, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (134):
- United States (134):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Beckman Research Institute, City of Hope, Duarte, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Van Nuys Breast Center, Van Nuys, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Hospital - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Ozarks Regional, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Hospital Tumor Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Badve SS, Baehner FL, Gray RP, Childs BH, Maddala T, Liu ML, Rowley SC, Shak S, Perez EA, Shulman LJ, Martino S, Davidson NE, Sledge GW, Goldstein LJ, Sparano JA. Estrogen- and progesterone-receptor status in ECOG 2197: comparison of immunohistochemistry by local and central laboratories and quantitative reverse transcription polymerase chain reaction by central laboratory. J Clin Oncol. 2008 May 20;26(15):2473-81. doi: 10.1200/JCO.2007.13.6424. PMID 18487567
- [Result] Goldstein LJ, Gray R, Badve S, Childs BH, Yoshizawa C, Rowley S, Shak S, Baehner FL, Ravdin PM, Davidson NE, Sledge GW Jr, Perez EA, Shulman LN, Martino S, Sparano JA. Prognostic utility of the 21-gene assay in hormone receptor-positive operable breast cancer compared with classical clinicopathologic features. J Clin Oncol. 2008 Sep 1;26(25):4063-71. doi: 10.1200/JCO.2007.14.4501. Epub 2008 Aug 4. PMID 18678838
- [Result] Goldstein LJ, Gray R, Childs BH, et al.: Prognostic utility of 21-gene assay in hormone receptor (HR) positive operable breast cancer and 0-3 positive axillary nodes treated with adjuvant chemohormonal therapy (CHT): an analysis of Intergroup trial E2197. [Abstract] J Clin Oncol 25 (Suppl 18): A-526, 2007.
- [Result] Goldstein LJ, O'Neill A, Sparano J, et al.: E2197: Phase III AT (doxorubucin/docetaxel) vs. AC (doxorubicin/cyclophosphamide) in the adjuvant treatment of node positive and high risk node negative breast cancer. [Abstract] J Clin Oncol 23 (Suppl 16): A-512, 7s, 2005.
- [Result] Goldstein LJ, O'Neill A, Sparano JA, et al.: LVEF assessment of adjuvant doxorubicin/cyclophosphamide (AC) vs. doxorubicin/docetaxel (AT) in early stage breast cancer: cardiac safety results of ECOG 2197. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-73, 2003.
- [Result] Goldstein L, Ravdin P, Gray R, et al.: Prognostic utility of the 21-gene assay compared with adjuvant in hormone receptor (HR) positive operable breast cancer with 0-3 positive axillary nodes treated with adjuvant chemohormonal therapy (CHT): an analysis of intergroup trial E2197. [Abstract] Breast Cancer Res Treat 106 (1): A-63, S17, 2007.
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/